CLINICAL TRIAL: NCT03459027
Title: Nitric Oxide Bioavailability and Dynamics of Blood Flow and Vasodilation With Age
Brief Title: Nitrate Supplementation and Muscle Blood Flow
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Iowa (Other)
Responsible Party: Principal Investigator, Darren P Casey, Assistant Professor, University of Iowa
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: 201708795
Record Dates: First submitted 2017-10-11; First posted 2018-03-08 (Actual); Last update posted 2019-01-09 (Actual); Status verified 2019-01

CONDITIONS: Vasodilation; Blood Pressure; Active Hyperemia; Aging
Keywords: exercise hyperemia; vasodilation; nitric oxide; dietary nitrate
MeSH Terms: conditions — Aneurysm; Hyperemia

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Nitrate Rich Beetroot Powder (nitrate) (Active Comparator): Dietary nitrate in the form of beetroot powder (10g) mixed in water will be administered acutely
  Interventions: Dietary Supplement: Super Beets; Dietary Supplement: Beetroot powder
- Placebo Beetroot Powder (Placebo Comparator): Beetroot powder devoid of nitrate (10g) will be mixed in water and administered acutely
  Interventions: Dietary Supplement: Super Beets; Dietary Supplement: Beetroot powder

INTERVENTIONS:
Dietary Supplement: Super Beets — Nitrate rich beetroot powder (10g) acutely
Dietary Supplement: Beetroot powder — Nitrate devoid beetroot powder (10g) acutely

SUMMARY:
The main purpose of this study is to evaluate the effects of an acute dose of dietary nitrate in the form of beetroot juice on skeletal muscle blood flow in response to dynamic knee extension exercise in healthy older adults. All subjects will receive active (rich in dietary nitrate) or placebo (devoid of nitrate) supplementation.

DETAILED DESCRIPTION:
Dietary nitrate (beetroot juice) is reduced to nitrite and nitric oxide within the digestive system of humans. Nitric oxide exerts potent vasodilator effects, which have been shown to reduce blood pressure and enhance exercise economy in humans. This pressure reducing effect may have implications within the regulation of blood flow during dynamic exercise in older adults.

ELIGIBILITY:
Inclusion Criteria:

* Healthy older adults 60-80 years of age

Exclusion Criteria:

* Hypertension,
* Smoking,
* Heart disease,
* Diabetes,
* Body mass index (BMI) ≥ 30 kg/m2,
* Autonomic disorders and other conditions that may alter blood pressure or vascular function
* Medications that might normally alter blood pressure or vascular function.
* Older women taking hormone replacement therapy medications.

Ages: 60 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2017-10-10 (Actual); Primary Completion 2018-02-08 (Actual); Study Completion 2018-02-08 (Actual)

PRIMARY OUTCOMES:
Change in Skeletal Muscle Blood Flow within the Leg via Doppler Ultrasound | Pre and 2 hours post acute ingestion of dietary nitrate and placebo with at least 5 days of separation between visits.
  Leg blood flow via Doppler ultrasound examined during dynamic knee extension exercise. Change in blood flow in response to dynamic knee exercise will be measured to examine the influence of dietary nitrate.

CONTACTS AND LOCATIONS:
Locations (1):
- Medical Education Building, Iowa City, Iowa, United States